CLINICAL TRIAL: NCT00648635
Title: A Pilot Study for Prospective Discovery of Possible Relationship Between Quality of Life, Treatment Modalities, and Patient Treatment/Outcome Expectations in Patients Undergoing Treatment for Locally Recurrent Rectal Adenocarcinoma
Brief Title: Relationship Between Quality of Life, Treatment Modalities, and Patient Treatment/Outcome Expectations
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0322; NCI-2020-07464 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Recurrent Rectal Adenocarcinoma; Quality of Life; QOL; Questionnaire; Survey
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PET + QOL: Survey of how recurrent rectal cancer treatment affects well being + QOL
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires taking 30-60 minutes to complete every 3 months.
  Other Names: Survey

SUMMARY:
The goal of this study is to learn how the treatment given to patients with recurrent rectal cancer affects their well being and quality of life.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete 4 questionnaires at each of your regularly scheduled doctor's visits (about every 6 months). Someone will help you to go through the questionnaires when you are given your first packet. If you are unable to complete the questionnaires while at your study visit, you may choose to take some or all of the questionnaires home. If you take the questionnaires home, you will be given a self-addressed stamped envelope so that you can return them to the study coordinator. If you choose, you may also complete the questionnaires over the phone.

The questionnaires will ask you about how you feel about the cancer treatment, how treatment for rectal cancer has affected your health and lifestyle, what you expect during and after your treatment, and about any pain you are experiencing and if the pain management is working for you. It should take about 30-60 minutes to complete the questionnaires each time.

If you will not be in the clinic for more than 6 months, the questionnaires will be mailed to you. You will return them in a self-addressed stamped envelope. If you have not completed the questionnaires within 2 weeks of receiving them, a research staff member will call you to remind you to complete the questionnaires, and to assist you with completing them (if necessary). If you have not completed the questionnaires by the time you come for your next follow-up visit, a research staff member will assist you with completing them at your visit (if necessary).

If your questionnaire responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive mental health screening.

At each of your appointments or between your appointments (if needed) researchers will collect study related information for your medical record.

Researchers will also review the images of the positron emission tomography (PET) scans or other diagnostic tests that you take as part of your standard of care. By viewing PET scan images or diagnostic tests, researchers hope to be able to discover whether there is any connection between the images on the PET scan or diagnostic tests and the symptoms that you are having. The PET scan or other diagnostic tests is are part of your standard treatment for your recurrent rectal cancer, and you will not have to have any special tests or scans just to participate in this study.

The data researchers collect will also be used to form a database of patients with recurrent rectal cancer. The database will be located on a password protected Surgical Oncology computer and it will be available only to the study doctor and the research staff that need to complete the study. The database will include information about each participant on the study. It will include information about the participant's name, medical record number, age, gender, diagnosis, the study questionnaires, and information about the disease.

Length of Study:

You will remain on study for up to 5 years.

This is an investigational study.

Up to 164 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who have had previous surgical treatment of rectal adenocarcinoma, regardless of age, with locally recurrent (pelvic) rectal adenocarcinoma are eligible, if a period of at least 3 months exists between initial treatment and disease recurrence.
2. Patients may have local recurrence alone, or concurrent distant metastatic disease. Patients must have recurrent rectal cancer present in the bony pelvis.
3. Patients must be conversant in English in order to complete appropriate questions.
4. Patients must understand the test and questionnaire parameters, including the need for PET testing to assess the correlation between perceived symptoms and PET or other diagnostic results. Patients must be able and willing to complete all scheduled appointments and complete and return all study questionnaires.

Exclusion Criteria:

1. Patients must not have non-adenocarcinoma pathology, i.e., squamous cell carcinoma of the anus, cloacogenic tumors, etc.
2. Patients must not have any concurrent pelvic malignancy in addition to rectal carcinoma.
3. Patients must not have ONLY distant metastases. Recurrence must be present within the bony pelvis.
4. Patients must not have a history of either a documented pelvic pain syndrome or a preoperative documented diagnosis of chronic constipation (defined as < 1 BM per 48 hours, unrelated to rectal cancer or mechanical obstruction) preceding the cancer diagnosis.
5. Patient must not have had solely non-operative therapies in treatment of their primary rectal carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with recurrent rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2008-03-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QOL) Survey Responses | Baseline and QOL at 6-month intervals for 5 years
  Primary endpoint of QOL assessed using EORTC QLQ-CR29 survey form. Change of QOL defined as the difference between the baseline and the QOL at 6-month intervals.

CONTACTS AND LOCATIONS:
Overall Officials: George J Chang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org